CLINICAL TRIAL: NCT00364897
Title: Comparison Between Two Tibial Fixation Techniques in ACL Reconstruction
Brief Title: Investigation of Clinical Outcome of ACL Reconstruction Utilizing Two Tibial Fixation Techniques, Concentric Tapered Interference Screws and Interference Screw and Sheath
Status: Withdrawn | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Other Study IDs: ACL001-HMO-CTIL
Record Dates: First submitted 2006-08-15; First posted 2006-08-16 (Estimated); Last update posted 2007-04-11 (Estimated); Status verified 2007-02

CONDITIONS: Primary ACL Tears

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
Tibial fixation is the weak link when using soft tissue grafts and interference screws for fixation in a bony tunnel in ACL reconstruction. The Objective is to study two groups of patients undergoing double loop hamstring autograft ACL reconstruction and compare between the two tibial fixation devices: the tapered Deltascrew and the Intrafix screw and sheath .

ELIGIBILITY:
Inclusion Criteria:

* Males and females between ages 21 and 40 years.
* Primary ACL tears.
* Signed Informed consent.
* Availability during follow up period.

Exclusion Criteria:

* Additional meniscal injury requiring suture.
* Articular cartilage injury requiring surgical management.
* Concomitant ligament injuries to the same knee requiring surgery.
* Bilateral ACL injury.
* Revision ACL surgery.
* Concurrent fractures of the lower limbs caused by the same accident.
* Post operative wound infection.

  • Post operative nerve injury
* Cardiovascular compromise.
* Professional sports people.
* Soldiers on active military service.
* Patients actively seeking compensation for injury.
* Patients on other research protocols.
* Patients receiving medications which alter bone metabolism: corticosteriods, Calcitonin, Flourides, Biphosphonates, Vitamin D and its derivatives, Cytotoxic drugs.
* Non compliance. • Pregnancy

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Lowe, Dr., Principal Investigator — Hadassah Medical Organization